CLINICAL TRIAL: NCT07142369
Title: Does Arthrocentesis and PRP For Acute ACL Tears With Hemarthrosis Decrease Inflammatory Cytokines At Time Of Surgery: A Prospective Randomized Control Trial (RCT)
Brief Title: Synovial Fluid Withdrawal or PRP Injection For Acute ACL Tears and Cytokines
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Arthroscopy Association of North America (AANA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24120505
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Posttraumatic Osteoarthritis; Anterior Cruciate Ligament (ACL) Rupture
Keywords: osteoarthritis
MeSH Terms: conditions — Rupture; Osteoarthritis | interventions — Arthrocentesis; Injections

STUDY DESIGN:
Intervention Model Description: Randomized control trial 1:1:1 study assignment (33 subjects Arm 1 two arthrocentesis withdrawals; 33 subjects Arm 2 two arthrocentesis withdrawals with PRP injection; 33 subjects Arm 3 a very small arthocentesis withdrawal and one standard arthrocentesis withdrawal and no PRP injection)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Two Synovial Fluid Withdrawals (Active Comparator): Subjects randomized to Arm 1 will have 2 synovial fluid withdrawals; one at the preoperative clinic visit and one at the time of surgery
  Interventions: Procedure: Synovial Fluid withdrawal at the preoperative clinic visit; Procedure: Synovial fluid withdrawal at the time of surgery
- Platelet-Rich Plasma (PRP) and Two Synovial Fluid Withdrawals (Experimental): Subjects randomized to ARM 2 will have 2 synovial fluid withdrawals one at the preoperative visit and one at the time of surgery. Platelet-Rich Plasma (PRP) preparation and injection will happen at the preoperative clinic visit.
  Interventions: Procedure: Synovial Fluid withdrawal at the preoperative clinic visit; Procedure: Platelet-Rich Plasma (PRP) preparation and injection; Procedure: Synovial fluid withdrawal at the time of surgery
- 3mL Synovial Fluid Withdrawal and Synovial Fluid Withdrawal at the Time of Surgery (Other): Subjects randomized to Arm 3 will have 3mL withdrawal of synovial fluid at the preoperative visit and 1 synovial fluid withdrawal at the time of surgery
  Interventions: Procedure: Synovial fluid withdrawal at the time of surgery; Procedure: 3mL synovial fluid withdrawn at the preoperative visit

INTERVENTIONS:
Procedure: Synovial Fluid withdrawal at the preoperative clinic visit — Synovial Fluid withdrawal at the preoperative clinic visit
  Other Names: arthrocentesis
  Arms: Platelet-Rich Plasma (PRP) and Two Synovial Fluid Withdrawals; Two Synovial Fluid Withdrawals
Procedure: Platelet-Rich Plasma (PRP) preparation and injection — Platelet-Rich Plasma (PRP) preparation and injection
  Other Names: platelet rich plasma
  Arms: Platelet-Rich Plasma (PRP) and Two Synovial Fluid Withdrawals
Procedure: Synovial fluid withdrawal at the time of surgery — Synovial fluid withdrawal at the time of surgery
Procedure: 3mL synovial fluid withdrawn at the preoperative visit — 3mL synovial fluid withdrawn at the preoperative visit
  Arms: 3mL Synovial Fluid Withdrawal and Synovial Fluid Withdrawal at the Time of Surgery

SUMMARY:
The purpose of this study is to determine what effects the withdrawal of excess knee joint fluid or the injection of a factor from the blood has on swelling after a sudden anterior cruciate ligament (ACL) rupture of the knee.

DETAILED DESCRIPTION:
The body responds to different stresses by releasing factors in the blood and fluids in response to stressors like injury, surgery or certain treatments. Some of these factors help heal and some make the injury and body swell (inflammation). In this study we want to see if the intervention of withdrawing fluid the knee or the addition of an enriched healing factor called platelet rich plasma (PRP) injected in the knee influences the body to produce healing factors in the knee joint fluid.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 50
* English-speaking
* Clinical evidence of ACL rupture with swelling
* Participant must be undergoing ACL reconstruction surgery

Exclusion Criteria:

* Age <18 or >50
* Presentation >3 weeks after initial injury
* Previous traumatic ipsilateral (same side) knee injury consistent with chronic ACL tear or prior ACL surgery
* > Kellgren-Lawrence grade 2 changes on preoperative x-ray
* History of hemophilia or inflammatory arthropathy (e.g., rheumatoid arthritis)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of Collagen Type II Cytokine | Enrollment up to surgery
  Breakdown cytokine found in damaged cartilage

CONTACTS AND LOCATIONS:
Overall Officials: Adam Yanke, MD, PhD, Principal Investigator — Associate Professor and Surgeon
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States